CLINICAL TRIAL: NCT05370157
Title: Improving Teamwork in Rural Child Advocacy Centers: A Hybrid-Effectiveness Implementation Trial of TeamTRACS
Brief Title: TeamTRACS Pilot (CTSI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Elizabeth McGuier, Assistant Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY21110090; UL1TR001857 (NIH)
Record Dates: First submitted 2022-04-26; First posted 2022-05-11 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Teamwork; Implementation
Keywords: multidisciplinary teamwork; implementation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) (Experimental): CACs randomized to the intervention condition (n = 4) will participate in TeamTRACS. CACs will receive an implementation guide to assist in preparing for and maximizing the impact of training.
  Interventions: Behavioral: TeamTRACS
- Waitlist Comparison (No Intervention): CACs randomized to the waitlist comparison (n = 2) will participate in TeamTRACS approximately 4 months after CACs in the intervention condition.

INTERVENTIONS:
Behavioral: TeamTRACS — TeamTRACS is a team training intervention adapted from TeamSTEPPS (Team Strategies and Tools to Enhance Performance and Patient Safety), a widely used evidence-based team training developed by the Agency for Healthcare Research and Quality. TeamTRACS targets knowledge, skills, and attitudes related to team member roles, shared awareness, communication, mutual support, and goal-setting. TeamTRACS is structured, easy to use, flexible in length and intensity, and requires few resources. It incorporates didactic instruction, discussion, and interactive activities and can be delivered virtually or in-person.
  Arms: TeamTRACS (Team Training in Roles, Awareness, Communication, and Support)

SUMMARY:
In a previous research study, the investigators adapted an evidence-based team training intervention for healthcare settings (TeamSTEPPS) to fit the needs and context of Child Advocacy Center multidisciplinary teams. This study is a cluster-randomized controlled trial of the adapted training, TeamTRACS (Team Training in Roles, Awareness, Communication, and Support). This hybrid type 2 effectiveness-implementation study will test the effectiveness of TeamTRACS and pilot a self-guided approach to implementing TeamTRACS in low-resource settings.

DETAILED DESCRIPTION:
This study is designed to test the effects of TeamTRACS on knowledge, skill use, and team functioning. It will also evaluate the acceptability, appropriateness, and feasibility of a self-guided implementation approach that requires few resources and builds local capacity for change. Six rural Child Advocacy Centers (CACs) will be randomized to TeamTRACS (4 CACs) or a waitlist comparison (2 CACs). The long-term goal of this research is to create an effective team training that can be rapidly scaled up and disseminated to rural CACs nationwide. Supporting rural teams can improve team performance, strengthen the workforce, and ultimately improve service quality and outcomes for rural children who experience child abuse.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 18 years of age who are members of the multidisciplinary team at the participating CACs.

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A McGuier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available upon reasonable request as allowed by IRB regulations and after manuscripts reporting the main findings are accepted for publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after manuscripts reporting the main findings are accepted for publication.
Access Criteria: Contact the principal investigator to request access to the deidentified data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only current team members were eligible to participate at each timepoint. Participants who completed baseline data collection but left the team before follow-up were not invited to participate in follow-up data collection. Participants who joined the team after baseline were invited to participate in follow-up data collection.
Units Other Than Participants: Children's Advocacy Centers
Period: Participants Entering at Baseline
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Started | 100; 4 Children's Advocacy Centers | 50; 2 Children's Advocacy Centers
Completed Baseline | 87; 4 Children's Advocacy Centers | 48; 2 Children's Advocacy Centers
Started Followup | 83; 4 Children's Advocacy Centers | 46; 2 Children's Advocacy Centers
Completed | 72; 4 Children's Advocacy Centers | 35; 2 Children's Advocacy Centers
Not Completed | 28; 0 Children's Advocacy Centers | 15; 0 Children's Advocacy Centers
Not completed — Lost to Follow-up | 11 | 11
Not completed — Not eligible for followup - no longer member of team | 17 | 4
Period: Participants Entering at Follow-Up
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Started (Participants who were not part of the team at baseline. All new participants were affiliated with participating Children's Advocacy Centers; no centers entered at follow-up.) | 17; 4 Children's Advocacy Centers | 5; 2 Children's Advocacy Centers
Completed | 17; 4 Children's Advocacy Centers | 5; 2 Children's Advocacy Centers
Not Completed | 0; 0 Children's Advocacy Centers | 0; 0 Children's Advocacy Centers

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for all unique participants
Groups:
- Total: Total of all reporting groups
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison | Total
Number analyzed (Participants) | 117 | 55 | 172
Age, Categorical [Count of Participants; unit: Participants] — Population: Age category is unknown for 13 participants
  Participants
    number analyzed (Participants) | 107 | 52 | 159
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 106 | 50 | 156
    >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age is unknown for 15 participants
  years
    number analyzed (Participants) | 105 | 52 | 157
    (all) | 39.46 (11.41) | 45.33 (11.46) | 41.40 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported Gender Population: Gender is unknown for 13 participants.
  Participants
    number analyzed (Participants) | 107 | 52 | 159
    Female | 74 | 39 | 113
    Male | 33 | 13 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 0 | 12
  Not Hispanic or Latino | 94 | 51 | 145
  Unknown or Not Reported | 11 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 0 | 12
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 8 | 9
  White | 92 | 43 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 117 | 55 | 172

OUTCOME MEASURES:

1. Primary Outcome: Change in Teamwork Knowledge From Baseline to 3-month Follow-up
Description: Survey questions assessing knowledge taught in TeamTRACS will be assessed with multiple choice questions. The percent of correct answers (range 0-100%) will be calculated.
Time Frame: Baseline, 3-month follow-up (Month 7, 3 months after training workshop)
Population: Descriptive data: Team members with data for that timepoint. Intent-to-treat analysis: All team members with data at 1 or more timepoints
Measure: Mean (Standard Deviation); unit: percentage correct answers
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Number analyzed (Participants) | 112 | 53
percentage correct answers
  Baseline: number analyzed (Participants) | 84 | 45
  Baseline | 75.60 (10.87) | 74.72 (10.82)
  Follow-up: number analyzed (Participants) | 85 | 40
  Follow-up | 80.00 (11.16) | 75.00 (7.88)
Statistical Analysis 1: Comparison: TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) vs Waitlist Comparison; Intent-to-treat analyses tested changes in knowledge from baseline to follow-up using linear mixed models. Mixed models analyses were conducted in R using the lme4 package and restricted maximum likelihood estimation (REML). Models included fixed effects of time (baseline vs. follow-up), intervention condition, and their interaction as well as random effects for person and team. We used the clubSandwich package to calculate cluster robust standard errors; Test type: Superiority; p = .03, Regression, Linear; Satterthwaite Approximation; Mean Difference (Net) = 4.25, 95% CI 2-sided [0.76 to 7.74], Standard Error of Mean 0.85

2. Primary Outcome: Change in Teamwork Skill Use From Baseline to 3-month Follow-up
Description: Frequency of teamwork skill use will be assessed with survey items rated on a 5-point Likert scale (range 1-5). Scores will be averaged; higher scores indicate more frequent skill use.
Time Frame: Baseline, 3-month follow-up (Month 7, 3 months after training workshop)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Number analyzed (Participants) | 111 | 52
score on a scale
  Baseline: number analyzed (Participants) | 83 | 44
  Baseline | 4.22 (0.49) | 4.08 (0.59)
  Follow-up: number analyzed (Participants) | 85 | 40
  Follow-up | 4.19 (0.54) | 4.20 (0.55)
Statistical Analysis 1: Comparison: TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) vs Waitlist Comparison; Intent-to-treat analyses tested changes in skill use from baseline to follow-up using linear mixed models. Mixed models analyses were conducted in R using the lme4 package and restricted maximum likelihood estimation (REML). Models included fixed effects of time (baseline vs. follow-up), intervention condition, and their interaction as well as random effects for person and team. We used the clubSandwich package to calculate cluster robust standard errors; Test type: Superiority; p = .30, Regression, Linear; Satterthwaite Approximation; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.40 to 0.20], Standard Error of Mean 0.08

3. Primary Outcome: Acceptability of Self-guided Implementation
Description: Perceived acceptability of the self-guided implementation process will be assessed with items from the Acceptability of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions.
Time Frame: Beginning, midpoint, and end of self-guided implementation process (Months 0, 5, & 7)
Population: Only rated by key informants in CACs randomized to TeamTRACS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Number analyzed (Participants) | 4 | 0
score on a scale
  Baseline (Beginning of self-guided implementation process) | 4.38 (0.48) |
  Month 5 (midpoint of self-guided implementation process) | 4.25 (0.96) |
  Month 7 (End of study) | 4.25 (0.50) |

4. Primary Outcome: Appropriateness of Self-guided Implementation
Description: Perceived appropriateness of the self-guided implementation process will be assessed with items from the Intervention Appropriateness Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions.
Time Frame: Beginning, midpoint, and end of self-guided implementation process (Months 0, 5, & 7)
Population: Only rated by key informants in CACs randomized to TeamTRACS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Number analyzed (Participants) | 4 | 0
score on a scale
  Baseline (Beginning of self-guided implementation process) | 3.63 (0.75) |
  Month 5 (midpoint of self-guided implementation process) | 4.25 (1.50) |
  Month 7 (End of study) | 4.25 (0.96) |

5. Primary Outcome: Feasibility of Self-guided Implementation
Description: Perceived feasibility of the self-guided implementation process will be assessed with items from the Feasibility of Intervention Measure. Each item is rated on a 1-5 Likert scale. Scores will be averaged; higher scores indicate more positive perceptions.
Time Frame: Beginning, midpoint, and end of self-guided implementation process (Months 0, 5, & 7)
Population: Only rated by key informants in CACs randomized to TeamTRACS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Number analyzed (Participants) | 4 | 0
score on a scale
  Baseline (Beginning of self-guided implementation process) | 4.50 (0.58) |
  Month 5 (midpoint of self-guided implementation process) | 4.00 (0.82) |
  Month 7 (End of study) | 4.38 (0.75) |

6. Secondary Outcome: Change in Team Functioning From Baseline to 3-month Follow-up: Psychological Safety
Description: Psychological safety (affective state) was assessed with Edmondson's (1999) Psychological Safety scale of 7 items rated on a 7-point Likert scale (1-7). Scores were averaged; higher scores indicate more psychological safety.
Time Frame: Baseline, 3-month follow-up (Month 7, 3 months after training workshop)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Number analyzed (Participants) | 111 | 52
score on a scale
  Baseline: number analyzed (Participants) | 82 | 44
  Baseline | 5.46 (1.12) | 5.59 (1.04)
  Follow-up: number analyzed (Participants) | 86 | 40
  Follow-up | 5.51 (1.13) | 5.94 (0.98)
Statistical Analysis 1: Comparison: TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) vs Waitlist Comparison; Intent-to-treat analyses tested changes in psychological safety from baseline to follow-up using linear mixed models. Mixed models analyses were conducted in R using the lme4 package and restricted maximum likelihood estimation (REML). Models included fixed effects of time (baseline vs. follow-up), intervention condition, and their interaction as well as random effects for person and team. We used the clubSandwich package to calculate cluster robust standard errors; Test type: Superiority; p = .45, Regression, Linear; Mean Difference (Net) = -0.23, 95% CI 2-sided [-1.25 to 0.79], Standard Error of Mean 0.25

7. Secondary Outcome: Change in Team Functioning From Baseline to 3-month Follow-up: Learning Behavior
Description: Learning behavior (behavioral process) was assessed with Edmondson's (1999) Learning Behavior scale of 7 items rated on a 7-point Likert scale (1-7). Scores were averaged; higher scores indicate more learning behavior.
Time Frame: Baseline, 3-month follow-up (Month 7, 3 months after training workshop)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Number analyzed (Participants) | 111 | 52
score on a scale
  Baseline: number analyzed (Participants) | 82 | 44
  Baseline | 4.77 (1.02) | 4.96 (1.02)
  Follow-up: number analyzed (Participants) | 86 | 40
  Follow-up | 4.86 (0.99) | 5.08 (0.96)
Statistical Analysis 1: Comparison: TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) vs Waitlist Comparison; Intent-to-treat analyses tested changes in learning behavior from baseline to follow-up using linear mixed models. Mixed models analyses were conducted in R using the lme4 package and restricted maximum likelihood estimation (REML). Models included fixed effects of time (baseline vs. follow-up), intervention condition, and their interaction as well as random effects for person and team. We used the clubSandwich package to calculate cluster robust standard errors; Test type: Superiority; p = .89, Regression, Linear; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.44 to 0.40], Standard Error of Mean 0.10

8. Secondary Outcome: Change in Team Performance From Baseline to 3-month Follow-up
Description: The overall quality of work done by the team will be assessed with Edmondson's (1999) Team Performance scale of 5 items rated on a 7-point Likert scale. Scores will be averaged; higher scores indicate better performance.
Time Frame: Baseline, 3-month follow-up (Month 7, 3 months after training workshop)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
Number analyzed (Participants) | 111 | 52
score on a scale
  Baseline: number analyzed (Participants) | 82 | 44
  Baseline | 5.47 (1.28) | 5.75 (1.08)
  Follow-up: number analyzed (Participants) | 86 | 40
  Follow-up | 5.63 (1.14) | 6.07 (0.97)
Statistical Analysis 1: Comparison: TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) vs Waitlist Comparison; Intent-to-treat analyses tested changes in team performance from baseline to follow-up using linear mixed models. Mixed models analyses were conducted in R using the lme4 package and restricted maximum likelihood estimation (REML). Models included fixed effects of time (baseline vs. follow-up), intervention condition, and their interaction as well as random effects for person and team. We used the clubSandwich package to calculate cluster robust standard errors; Test type: Superiority; p = .85, Regression, Linear; Mean Difference (Net) = -0.08, 95% CI 2-sided [-1.51 to 1.36], Standard Error of Mean 0.36

ADVERSE EVENTS:
Time Frame: Up to 9 months
Description: All-Cause Mortality among participants was not assessed; therefore the number of participants at risk for All-Cause Mortality is zero.
Arm/Group | TeamTRACS (Team Training in Roles, Awareness, Communication, and Support) | Waitlist Comparison
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/55
Other Adverse Events (participants affected / at risk) | 0/117 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT05370157/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT05370157/ICF_000.pdf